CLINICAL TRIAL: NCT06049719
Title: Translation, Cross-cultural Adaptation and Validation of the Turkish Version of NIH Task Force's Recommended Multidimensional Minimal Dataset for Research on Chronic Low Back Pain
Brief Title: Reliabılıty,Validity Of The Turkish Version Of The NIH-Minimal Dataset
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, GÖKHAN MARAŞ, Research assistant, Gazi University
Other Study IDs: 2022-18-2
Record Dates: First submitted 2023-09-13; First posted 2023-09-22 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: validity; reliability; low back apain; translation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Patients with low back pain (18-65 years)
  Interventions: Other: NIH Task Force's Recommended Multidimensional Minimal Dataset

INTERVENTIONS:
Other: NIH Task Force's Recommended Multidimensional Minimal Dataset — Questionnaire
  Other Names: Turkish version of the NIH Task Force's Recommended Multidimensional Minimal Dataset

SUMMARY:
This study, we performed the Turkish version validity and reliability of the NIH Task Force's Recommended Multidimensional Minimal Dataset

DETAILED DESCRIPTION:
Low back pain is defined as the pain that can occur in the region between the lower border of the scapula and the hip, sometimes spreading to the lower extremities, which causes activity limitation and is one of the most common health problems in the society. Appropriate use of assessment questionnaires is one of the most important steps in the evaluation of the functional level of the patient and in deciding on an effective treatment protocol. The purpose of our study is to determine the Turkish version, validity and reliability of NIH Task Force's Recommended Multidimensional Minimal Dataset. 200 patients with chronic low back pain were included in the study. Test-retest and internal consistency analysis were conducted to determine the reliability of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Having a low back pain Literate

Exclusion Criteria:

* pregnant,
* canser
* trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with chronic low back pain.
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Roland Morris disability questionnaire | 10 minute
  Roland Morris Disability Questionnaire, a widely used health status measure for low back pain. The RMDQ can be used in research or clinical practice.
Oswestry Low Back Pain Disability Questionnaire | 10 minute
  The Oswestry Disability Index (ODI) has become one of the principal condition-specific outcome measures used in the management of spinal disorders

CONTACTS AND LOCATIONS:
Overall Officials: Seyit Citaker, Prof., Study Chair — Gazi University
Locations (3):
- Turkey (Türkiye) (3):
  - Gazi University, Ankara
  - Gokhan MARAS, Ankara
  - Gökhan maraş, Ankara

IPD SHARING:
Plan to Share IPD: Yes